CLINICAL TRIAL: NCT05532254
Title: A Randomized, Single Oral Dose, Two-way Crossover, Open-label, Laboratory Blind, Bioequivalence Study Comparing Aripiprazole From Two Different Drug Products After Oral Administration to Healthy Adult Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Aripiprazole in Healthy Adult Subjects Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, Hala Masoud, FRC Technical Director & CEO, Future University in Egypt
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: ARI-B-20-031
Record Dates: First submitted 2022-09-04; First posted 2022-09-08 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Healthy Subjects
Keywords: Bioequivalence; Randomized; Crossover; Aripiprazole
MeSH Terms: interventions — Aripiprazole; Tablets

STUDY DESIGN:
Intervention Model Description: A randomized, single-dose, two-way crossover, open-label, laboratory blind, bioequivalence study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Product (T) (Experimental): subjects were administered a single tablet of 10 mg Aripiprazole with approximately 240 ml water after an overnight fast of 10 hours
  Interventions: Drug: Aripiprazole 10 mg tablet
- Reference Product (R) (Active Comparator): subjects were administered a single tablet of 10 mg Aripiprazole with approximately 240 ml water after an overnight fast of 10 hours
  Interventions: Drug: Abilify® 10 mg tablet

INTERVENTIONS:
Drug: Aripiprazole 10 mg tablet — an immediate-release tablet containing 10 mg Aripiprazole
  Other Names: Test product (T)
  Arms: Test Product (T)
Drug: Abilify® 10 mg tablet — an immediate-release tablet containing 10 mg Aripiprazole
  Other Names: Reference product (R)
  Arms: Reference Product (R)

SUMMARY:
To evaluate and compare the relative plasma bioavailability and therefore the bioequivalence of two different immediate release products each containing Aripiprazole 10 mg, after administering a single oral dose, to healthy adult subjects under fasting conditions.

DETAILED DESCRIPTION:
Enrolled subjects were randomized in a two-phase, two-sequence, cross-over design to receive a single dose of the test product (T) or the reference product (R) at each phase, under fasting conditions, with a wash-out period of 21 days.

Aripiprazole plasma concentration was determined using a validated LC-MS-MS method, followed by Pharmacokinetics, and statistical analysis using Phoenix WinNonlin® software to determine the average bioequivalence.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained for the study.
* Age 35 - 55 years
* Body mass index between 18.5 and 30 kg/m2
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination.
* Vital signs without significant deviations.
* All laboratory screening results are within the normal range or clinically non-significant

Exclusion Criteria:

* History or presence of any disorder or condition that would render the subject unsuitable for the study, place the subject at undue risk or interfere with the ability of the subject to complete the study in the investigator's opinion.
* History of significant cardiovascular, hepatic, renal, respiratory, gastrointestinal, endocrine, immunologic, allergic, dermatologic, hematologic, neurologic, or psychiatric disease, or cancer.
* Any confirmed significant allergic reactions against any drug or multiple allergies.
* Clinically significant illness 28 days before study phase I.
* Alcohol or any solvent intake.
* Regular use of medication.
* Positive urine screening of drugs of abuse.
* Use any systemic medications (prescription medications, OTC products, supplements, or herbal preparations) for 14 days prior to dosing and during the study.
* History or presence of significant smoking (more than one pack per day of cigarettes) or refusal to abstain from smoking for 48 hours before dosing until checkout.
* Blood donation within the past 60 days.
* Participation in another bioequivalence study within 60 days prior to the start of phase I of the study.

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2021-02-14 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Pre-dose (0) and at 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 48, 72 hours post dose
  Cmax is observed as the maximum of Aripiprazole peak concentration
Truncated area under the plasma concentration curve from administration to last observed (AUC 0-72h) | Pre-dose (0) and at 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 48, 72 hours post dose
  The AUC (0-72h) is the area under the Aripiprazole plasma concentration with time curve from the time of dosing to the 72-hour sample

SECONDARY OUTCOMES:
Maximum time (Tmax) | Pre-dose (0) and at 0.5, 1, 1.5, 2, 2.5,3, 3.5, 4, 4.5, 5, 5.5, 6, 8, 10, 12, 24, 48, 72 hours post dose
  Time until Cmax is reached

CONTACTS AND LOCATIONS:
Overall Officials: Hala Masoud, PhD, Principal Investigator — Future Research Center (FRC)
Locations (1):
- Future Research Center (FRC), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this study, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months following article publication and no end date
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to <hala.fut.masoud@gmail.com> To gain access.